CLINICAL TRIAL: NCT01577160
Title: An Open Label, Prospective, Non-Comparative Study to Evaluate Flexible Dose of Paliperidone ER and Clinical Response in the Treatment of Subjects With Schizophrenia
Brief Title: A Study to Evaluate Flexible Dose of Paliperidone Extended Release (ER) and Clinical Response in Participants With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015664; R076477SCH4034 (Other: Johnson & Johnson Taiwan Ltd); PAL-TWN-MA2 (Other: Johnson & Johnson Taiwan Ltd)
Record Dates: First submitted 2012-04-12; First posted 2012-04-13 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Extended Release (ER)
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Extended Release (ER) (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Participants will receive paliperidone ER 6 milligram (mg) orally once daily up to Week 12. Dose adjustment will be done at Week 2, 4 and 8 as per investigator's discretion based upon participant's CGI-I score.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of paliperidone ER for the treatment of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) participants.

DETAILED DESCRIPTION:
This is a multi-center (when more than one hospital or medical school team work on a medical research study), open-label (all people know the identity of the intervention), prospective (study following participants forward in time), non-comparative study. The total study duration will be 12 weeks for each participant and will include following visits: Screening, Week 2, 4, 8, and 12 (end of treatment or early withdrawal). The effectiveness of paliperidone ER will be evaluated at Week 12 by the proportion of responders who are evaluated as "very much improved" or "much improved" on the Clinical Global Impression improvement (CGI-I) Scale. Participants' safety will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with schizophrenia (according to Diagnostic and Statistical Manual of Mental Disorders [Edition 4] criteria)
* Participants with Clinical Global Impression-Severity (CGI-S) score greater than or equal to 4 points (moderately ill) at Screening
* Childbearing potential women who consented to the consistent use of the acceptable contraception (oral contraceptive, contraceptive injection, intrauterine device, double barrier method and contraceptive patch)
* Participants who are capable of and willing to fill out the questionnaire for themselves
* Participants who are compliant with self-medication or can receive consistent help or support

Exclusion Criteria:

* Participants with the past history of neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness)
* Participants with allergy or hypersensitivity to risperidone or paliperidone
* Participants who have taken clozapine, or have been exposed to the study drug within one month before screening
* Participants who have been treated with the long acting antipsychotic injection within 28 days
* Participants with significant risk including suicide or aggressive behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan Ltd Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone ER: Participants received paliperidone ER 6 milligram (mg) orally once daily up to Week 12. Dose adjustment was done at Week 2, 4 and 8 as per Investigator's discretion based upon participant's Clinical Global Impression - Improvement (CGI-I) score.
Period: Overall Study
Arm/Group | Paliperidone ER
Started | 353
Completed | 255
Not Completed | 98
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 15
Not completed — Lost to Follow-up | 40
Not completed — Withdrawal by Subject | 18
Not completed — Subject Uncooperative | 7
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone ER: Participants received paliperidone ER 6 milligram (mg) orally once daily up to Week 12. Dose adjustment was done at Week 2, 4 and 8 as per Investigator's discretion based upon participant's CGI-I score.
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 221

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders as Per Clinical Global Impression - Improvement (CGI-I) Scale
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Responders were defined as participants evaluated as "1: very much improved" or "2: much improved" on the CGI-I scale at Week 12.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Here 'N' (Number of Participants Analyzed) signifies those participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paliperidone Extended Release (ER): Participants received paliperidone ER 6 milligram (mg) orally once daily up to Week 12. Dose adjustment was done at Week 2, 4 and 8 as per Investigator's discretion based upon participant's CGI-I score.
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 255
percentage of participants | 21.6 [16.68 to 27.13]

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 12
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, Week 12
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Here, 'n' signifies those participants who were evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 331
units on a scale
  Baseline (n=331) | 5.0 (0.8)
  Change at Week 12 (n=255) | -1.4 (1.0)

3. Secondary Outcome: Number of Participants With Clinical Global Impression - Improvement (CGI-I) Score
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Week 12
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Here 'N' (Number of Participants Analyzed) signifies those participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 255
participants
  Very much improved | 3 (0.9)
  Much improved | 52
  Minimally improved | 119
  No change | 67
  Minimally worse | 10
  Much worse | 2
  Very much worse | 2

4. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Score at Week 12
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 331
units on a scale
  Baseline (n=331) | 42.6 (14.9)
  Change at Week 12 (n=267) | 14.3 (13.0)

5. Secondary Outcome: Change From Baseline in Drug Attitude Inventory (DAI-10) Score at Week 12
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response (SR). A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive SR; a negative sum of scores indicates a negative SR (non-compliant). The final score is the grand total of the positive and negative points. Total score ranges from (-) 10 to (+) 10, higher score indicates positive SR (compliant) and lower score indicates negative SR (non-compliant).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 331
units on a scale
  Baseline (n=331) | 2.5 (4.6)
  Change at Week 12 (n=267) | 1.0 (4.9)

ADVERSE EVENTS:
Arm/Group | Paliperidone ER
Serious Adverse Events (participants affected / at risk) | 0/353
Other Adverse Events (participants affected / at risk) | 140/353
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=353)
Constipation (Gastrointestinal disorders) | 40
Pyrexia (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 18
Upper Respiratory Tract Infection (Infections and infestations) | 18
Wound (Injury, poisoning and procedural complications) | 9
Extrapyramidal Disorder (Nervous system disorders) | 34
Headache (Nervous system disorders) | 9
Anxiety (Psychiatric disorders) | 25
Delusion (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 56
Cough (Respiratory, thoracic and mediastinal disorders) | 13

LIMITATIONS AND CAVEATS:
Some Adverse Events summaries were reported based on estimates due to the fact that they were not prepared in the original study report and the relevant definitions of the data elements were not available for these summaries to be regenerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less